CLINICAL TRIAL: NCT02283762
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Study to Investigate the Efficacy and Safety of Riociguat in Patients With Diffuse Cutaneous Systemic Sclerosis (dcSSc)
Brief Title: Efficacy and Safety of Riociguat in Patients With Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16277; 2014-001353-16 (EudraCT Number)
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Riociguat (Experimental): Main treatment phase of 52 weeks: participants received increasing doses of riociguat by 0.5 mg every 2 weeks up to 2.5 mg 3 times a day (TID) in a-titration period of up to 10 weeks and a maintenance period of up to 42 weeks. Long-term extension phase: starting after the completion of the Main Treatment Phase in Week 52, participants received sham-titration in a dose-titration period of up to 10 weeks followed by a maintenance period.
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)
- Placebo (Placebo Comparator): Main treatment phase of 52 weeks: participants received matching placebo tablets to riociguat as sham titration in a dose-titration period up to 10 weeks and a maintenance period of up to 42 weeks. Long-term extension phase: starting after the completion of the Main Treatment Phase in Week 52, participants received increasing doses of riociguat by 0.5 mg every 2 weeks up to 2.5 mg 3 times a day (TID) in a dose-titration period of up to 10 weeks followed by a maintenance period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — Starting dose 0.5 mg TID, increase by 0.5 mg every 2 weeks until highest possible dose of 2.5 mg TID
  Arms: Riociguat
Drug: Placebo — Sham-titration
  Arms: Placebo

SUMMARY:
To investigate if Riociguat is effective in the treatment of systemic sclerosis

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years and older
* Systemic sclerosis, as defined by ACR/EULAR (American College of Rheumatology/European League Against Rheumatism) 2013 criteria
* dcSSc (diffuse cutaneous systemic sclerosis) according to the LeRoy criteria, ie, skin fibrosis proximal to the elbows and knees in addition to acral fibrosis
* Disease duration of ≤ 18 months (defined as time from the first non-Raynaud's phenomenon manifestation)
* ≥ 10 and ≤ 22 mRSS (modified Rodnan skin score) units at the screening visit
* FVC (forced vital capacity) ≥ 45% of predicted at screening
* DLCO (diffusion capacity of the lung for carbon monoxide) ≥ 40% of predicted (hemoglobin-corrected) at screening
* Negative serum pregnancy test in a woman of childbearing potential at the screening visit
* Women of childbearing potential must agree to use adequate contraception when sexually active. "Adequate contraception" is defined as any combination of at least 2 effective methods of birth control, of which at least 1 is a physical barrier (e.g. condom with hormonal contraception like implants or combined oral contraceptives, condom with intrauterine devices). This applies since signing of the informed consent form until 30 (+5) days after the last study drug administration.

Exclusion Criteria:

* Limited cutaneous SSc (systemic sclerosis) at screening
* Major surgery (including joint surgery) within 8 weeks prior to screening
* Hepatic insufficiency classified as Child-Pugh C
* Patients with isolated AST or ALT >3xULN or bilirubin >2xULN can be included in the trial under the condition of additional monitoring during the trial
* Estimated glomerular filtration rate (eGFR) < 15 mL/min/1.73 m^2 (Modification of Diet in Renal Disease formula) or on dialysis at the screening visit. Patients entering the trial with eGFR 15-29 mL/min/1.73 m^2 will be undergo additional monitoring of renal function
* Any prior history of renal crisis
* Sitting SBP (systolic blood pressure) < 95 mmHg at the screening visit
* Sitting heart rate < 50 beats per minute (BPM) at the screening visit
* Left ventricular ejection fraction < 40% prior to screening
* Any form of pulmonary hypertension as determined by right heart catheterization
* Pulmonary disease with FVC < 45% of predicted or DLCO (hemoglobin-corrected) < 40% of predicted at screening
* Active state of hemoptysis or pulmonary hemorrhage, including those events managed by bronchial artery embolization
* Not permitted prior and concomitant medication
* Pregnant or breast feeding women
* Women of childbearing potential not willing to use adequate contraception and not willing to agree to 4-weekly pregnancy testing from Visit 1 (first administration of study drug) onwards until 30 (+5) days after last study drug intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (59):
- United States (10):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Michigan Health System, Ann Arbor, Michigan
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Medical University of South Carolina Medical Center, Charleston, South Carolina
  - Memorial Hermann-Texas Medical Center, Houston, Texas
  - University of Utah Health Care, Salt Lake City, Utah
- Australia (5):
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital, Fitzroy, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (3):
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Canada (4):
  - St. Joseph's Healthcare - Hamilton, Hamilton, Ontario
  - Arthritis Program Research Group, Inc., Newmarket, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
- Revmatologicky ustav, Prague, Czechia
- France (5):
  - Hôpital Pellegrin - Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire - Grenoble, Grenoble
  - Hopital Claude-Huriez CHRU, Lille
  - Cochin - Paris, Paris
  - CHU STRASBOURG - Hôpital de Hautepierre, Strasbourg
- Germany (4):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Kerckhoff-Klinik GmbH, Bad Nauheim, Hesse
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
- Hungary (2):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Italy (5):
  - A.O.U. Policlinico Umberto I, Rome, Lazio
  - A.O.U. di Cagliari, Cagliari, Sardinia
  - A.O.U. Careggi, Florence, Tuscany
  - A.O.U. Pisana, Pisa, Tuscany
  - A.O. di Padova, Padua, Veneto
- Japan (5):
  - Gunma University Hospital, Maebashi, Gunma
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tohoku University Hospital, Sendai, Miyagi
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Institute of Rheumatology Tokyo Women's Medical University, Shinjuku-ku, Tokyo
- Netherlands (2):
  - Universitair Medisch Centrum St. Radboud, Nijmegen
  - University Medical Center Utrecht, Utrecht
- Wellington Hospital, Wellington, New Zealand
- Switzerland (3):
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Universitätsspital Basel, Basel
  - UniversitätsSpital Zürich, Zurich
- Turkey (Türkiye) (4):
  - Cukurova Univ. Tip. Fak. Balcali Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
- United Kingdom (5):
  - Hope Hospital, Salford, Manchester
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Ninewells Hospital, Dundee
  - Aintree University Hospital, Liverpool
  - Royal Free Hospital, London

REFERENCES:
- [Background] Distler O, Pope J, Denton C, Allanore Y, Matucci-Cerinic M, de Oliveira Pena J, Khanna D. RISE-SSc: Riociguat in diffuse cutaneous systemic sclerosis. Respir Med. 2017 Jan;122 Suppl 1:S14-S17. doi: 10.1016/j.rmed.2016.09.011. Epub 2016 Sep 28. PMID 27746061
- [Derived] Khanna D, Kramer F, Hofler J, Ghadessi M, Sandner P, Allanore Y, Denton CP, Kuwana M, Matucci-Cerinic M, Pope JE, Atsumi T, Becvar R, Czirjak L, De Langhe E, Hachulla E, Ishii T, Ishikawa O, Johnson SR, Riccieri V, Schiopu E, Silver RM, Smith V, Stagnaro C, Steen V, Stevens W, Szucs G, Truchetet ME, Wosnitza M, Distler O. Biomarker analysis from the phase 2b randomized placebo-controlled trial of riociguat in early diffuse cutaneous systemic sclerosis. Rheumatology (Oxford). 2024 Nov 1;63(11):3124-3134. doi: 10.1093/rheumatology/keae150. PMID 38460548
- [Derived] Distler O, Allanore Y, Denton CP, Kuwana M, Matucci-Cerinic M, Pope JE, Atsumi T, Becvar R, Czirjak L, Hachulla E, Ishii T, Ishikawa O, Johnson SR, De Langhe E, Stagnaro C, Riccieri V, Schiopu E, Silver RM, Smith V, Steen V, Stevens W, Szucs G, Truchetet ME, Wosnitza M, Laapas K, Kramer F, Khanna D. Riociguat in patients with early diffuse cutaneous systemic sclerosis (RISE-SSc): open-label, long-term extension of a phase 2b, randomised, placebo-controlled trial. Lancet Rheumatol. 2023 Nov;5(11):e660-e669. doi: 10.1016/S2665-9913(23)00238-2. PMID 38251533
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 15 January 2015 (first patient first visit) and 28 March 2019 (last patient last visit). The Main Treatment Phase has been conducted between 15 Jan 2015 (first subject first visit) and 03 Jan 2018 (last subject last visit for the main treatment phase).
Pre-assignment Details: 139 patients were screened in 60 study centers in 15 countries worldwide. 121 patients of 139 patients were randomized and treated with at least one dose of study medication.
  88 of the 121 randomized patients completed the treatment phase, of whom 87 entered the long term extension (LTE) phase.
Groups:
- Riociguat (Adempas, BAY63-2521): Main treatment phase of 52 weeks: participants received increasing doses of riociguat by 0.5 mg every 2 weeks up to 2.5 mg 3 times a day (TID) in a-titration period of up to 10 weeks and a maintenance period of up to 42 weeks. Long-term extension phase: starting after the completion of the Main Treatment Phase in Week 52, participants received sham-titration in a dose-titration period of up to 10 weeks followed by a maintenance period.
- Placebo: Main treatment phase of 52 weeks: participants received matching placebo tablets to riociguat as sham-titration in a dose-titration period up to 10 weeks and a maintenance period of up to 42 weeks. Long-term extension phase: starting after the completion of the Main Treatment Phase in Week 52, participants received increasing doses of riociguat by 0.5 mg every 2 weeks up to 2.5 mg 3 times a day (TID) in a dose-titration period of up to 10 weeks followed by a maintenance period.
Period: Main Treatment Phase (MT)
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Started | 60 | 61
Completed | 42 | 46
Not Completed | 18 | 15
Not completed — Adverse Event | 9 | 9
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 7 | 4
Period: Long-term Extension Phase (LTE)
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Started | 42 | 45 (Of the 46 patients who completed the main treatment phase, 1 patient did not enter the LTE phase)
Completed | 32 | 31
Not Completed | 10 | 14
Not completed — Adverse Event | 2 | 6
Not completed — Lack of Efficacy | 1 | 1
Not completed — Study terminated at site | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (11.5) | 49.5 (12.9) | 50.7 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 45 | 92
  Male | 13 | 16 | 29
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 43 | 46 | 89
  Black | 2 | 3 | 5
  Asian | 12 | 12 | 24
  Native Hawaiian or other pacific islander | 1 | 0 | 1
  Not Hispanic or Latino | 59 | 58 | 117
Modified Rodnan skin score (mRSS) [Mean (Standard Deviation); unit: score on a scale] — The mRSS is a validated physical examination method for estimating skin thickness. It correlates with biopsy measures of collagen in the dermis and reflects prognosis and visceral involvement, especially in early disease. It is scored on 0 (normal) to 3+ (severe induration) ordinal scales over 17 body areas, with a maximum score of 51 (higher score means worse situation) and is used to categorize severity of systemic sclerosis (SSc).
  score on a scale | 16.9 (3.4) | 16.7 (4.1) | 16.8 (3.7)
Forced vital capacity (FVC) percent predicted [Mean (Standard Deviation); unit: FVC percent predicted] — Pulmonary function tests included forced vital capacity (FVC) and diffusion capacity of the lung for carbon monoxide (DLCO). FVC percent predicted was reported.
  FVC percent predicted | 90.743 (18.523) | 94.823 (17.034) | 92.800 (17.832)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Rodnan Skin Score (mRSS) to Week 52
Description: The mRSS is a validated physical examination method for estimating skin thickness. It correlates with biopsy measures of collagen in the dermis and reflects prognosis and visceral involvement, especially in early disease. It is scored on 0 (normal) to 3+ (severe induration) ordinal scales over 17 body areas, with a maximum score of 51 (higher score means worse situation) and is used to categorize severity of SSc. A decrease in the mean change of mRSS shows mRSS improved.
Time Frame: Baseline to week 52
Population: Full analysis set (FAS: all participants randomized and treated with study medication) with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 57 | 52
score on a scale | -2.088 (5.658) | -0.769 (8.243)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) vs Placebo; Test type: Superiority; p = 0.0815, MMRM (Method 1); Difference of LS means = -2.34, 95% CI 2-sided [-4.99 to 0.30]

2. Secondary Outcome: CRISS (American College of Rheumatology Composite Response Index for Clinical Trials) at Week 52 Reported as Number of Participants With a CRISS Probability >=0.60 or <0.60 From Baseline to Week 52
Description: CRISS forms a composite response index consisting of SSc-related organ involvement and the following five variables: mRSS, FVC percent predicted, physician's and patient's global assessments, and HAQ-DI score (from SHAQ patient-reported outcome). The resulting index is a 2-step process that captures clinically meaningful worsening of internal organ involvement and the core variables that show change. Patients for whom the predicted CRISS probability was ≥ 0.60 were considered improved, while patients for whom the predicted probability was < 0.60 were considered not improved.
Time Frame: Week 52
Population: Full analysis set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 60 | 61
Participants
  CRISS probability ≥ 0.60 | 11 | 11
  CRISS probability < 0.60 | 49 | 50
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) vs Placebo; Test type: Superiority — The pre-specified test was for superiority but ONLY if the primary endpoint and secondary endpoints were meeting statistical significance (hierarchical testing); p = 0.9770, Mantel Haenszel; % = 0.2, 95% CI 2-sided [-13.68 to 14.09]

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score to Week 52
Description: The HAQ-DI is a composite measure from which a 'Standard Disability Index' score can be computed to assess a patient's disability level. Generally, a score of 0-1 represents mild to moderate difficulty, 1-2 moderate to severe disability and 2-3 severe to very severe disability. The HAQ-DI comprises 20 items that assess patient abilities across 8 functional activities: dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. Each item is rated on a 4-point scale: 0=Without ANY difficulty, 1=With SOME difficulty, 2=With MUCH difficulty, 3=UNABLE to do. The 8 scores of the 8 sections are summed and divided by 8. In the event that one section is not completed by a subject then the summed score would be divided by 7. The final overall HAQ-DI score ranges from 0 to 3 and positive change indicates worse health-related quality of life (HRQoL).
Time Frame: Baseline to week 52
Population: FAS with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 60 | 61
score on a scale
  Baseline | 0.888 (0.665) | 0.693 (0.688)
  Change from baseline: number analyzed (Participants) | 56 | 52
  Change from baseline | 0.054 (0.381) | 0.127 (0.418)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) vs Placebo; change from baseline; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.3529, MMRM (Method 1); Difference in LS means = -0.07, 95% CI 2-sided [-0.23 to 0.08]

4. Secondary Outcome: Change From Baseline in Patient's Global Assessment Score to Week 52
Description: The patient's global assessments (a self-report) quantified the overall disease activity or severity of SSc, with scores ranging from 0 (good) to 10 (worse). Positive change in the patient's global assessments score indicates worsening.
Time Frame: Baseline to week 52
Population: FAS with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 60 | 61
score on a scale
  Baseline | 3.933 (2.497) | 3.770 (2.341)
  Change from baseline: number analyzed (Participants) | 45 | 46
  Change from baseline | 0.689 (2.745) | -0.022 (2.226)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) vs Placebo; Change from baseline; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0887, MMRM (Method 1); Difference in LS means = 0.79, 95% CI 2-sided [-0.12 to 1.69]

5. Secondary Outcome: Change From Baseline in Physician's Global Assessment Score to Week 52
Description: The physician's global assessments (reported by the physician) quantified the overall disease activity or severity of SSc, with scores ranging from 0 (good) to 10 (worse). Positive change in the physician's global assessments score indicates worsening.
Time Frame: Baseline to week 52
Population: FAS with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 60 | 61
score on a scale
  Baseline | 4.333 (2.105) | 4.016 (2.004)
  Change from baseline: number analyzed (Participants) | 45 | 47
  Change from baseline | -0.067 (2.157) | -0.745 (2.090)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) vs Placebo; Change from baseline; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0241, MMRM (Method 1); Difference in LS means = 0.83, 95% CI 2-sided [0.11 to 1.54]

6. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) Percent Predicted to Week 52
Description: Negative change in FVC percent predicted indicates worsening.
Time Frame: Baseline to week 52
Population: FAS with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: FVC percent predicted
Arm/Group | Riociguat (Adempas, BAY63-2521) | Placebo
Number analyzed (Participants) | 55 | 51
FVC percent predicted | -2.376 (7.515) | -2.945 (9.727)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) vs Placebo; change from baseline; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.9010, MMRM (Method 1); Difference in LS means = -0.20, 95% CI 2-sided [-3.40 to 3.00]

ADVERSE EVENTS:
Time Frame: From first application of study drug up to 2 days after end of treatment with study drug, up to 4 years.
Description: All 42 patients who completed the main treatment phase from the riociguat group entered the LTE phase and continued to receive riociguat. This group is referred in the LTE phase to "riociguat-riociguat group". One of the 46 patients from the placebo group did not enter the LTE phase. This group is referred to "placebo-riociguat group".
Groups:
- Riociguat-Riociguat (LTE Phase): Main treatment phase: participants received increasing doses of riociguat by 0.5 mg every 2 weeks up to 2.5 mg 3 times a day (TID) in a-titration period of up to 10 weeks and a maintenance period of up to 42 weeks. Long-term extension phase: starting from Week 52, participants received sham-titration in a dose-titration period of up to 10 weeks followed by a maintenance period.
- Placebo-Riociguat (LTE Phase): Main treatment phase: participants received matching placebo tablets to riociguat as sham-titration in a dose-titration period up to 10 weeks and a maintenance period of up to 42 weeks. Long-term extension phase: starting from Week 52, participants received increasing doses of riociguat by 0.5 mg every 2 weeks up to 2.5 mg 3 times a day (TID) in a dose-titration period of up to 10 weeks followed by a maintenance period.
- Riociguat (Main Treatment Phase): Main treatment phase of 52 weeks: participants received increasing doses of riociguat by 0.5 mg every 2 weeks up to 2.5 mg 3 times a day (TID) in a-titration period of up to 10 weeks and a maintenance period of up to 42 weeks. Long-term extension phase: starting after the completion of the Main Treatment Phase in Week 52, participants received sham-titration in a dose-titration period of up to 10 weeks followed by a maintenance period.
- Placebo (Main Treatment Phase): Main treatment phase of 52 weeks: participants received matching placebo tablets to riociguat as sham-titration in a dose-titration period up to 10 weeks and a maintenance period of up to 42 weeks. Long-term extension phase: starting after the completion of the Main Treatment Phase in Week 52, participants received increasing doses of riociguat by 0.5 mg every 2 weeks up to 2.5 mg 3 times a day (TID) in a dose-titration period of up to 10 weeks followed by a maintenance period.
Arm/Group | Riociguat-Riociguat (LTE Phase) | Placebo-Riociguat (LTE Phase) | Riociguat (Main Treatment Phase) | Placebo (Main Treatment Phase)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/45 | 1/60 | 1/61
Serious Adverse Events (participants affected / at risk) | 10/42 | 11/45 | 9/60 | 15/61
Other Adverse Events (participants affected / at risk) | 38/42 | 39/45 | 55/60 | 49/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat-Riociguat (LTE Phase) (N=42) | Placebo-Riociguat (LTE Phase) (N=45) | Riociguat (Main Treatment Phase) (N=60) | Placebo (Main Treatment Phase) (N=61)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scleroderma renal crisis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Prophylaxis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salpingitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site joint infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ultrasound kidney abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat-Riociguat (LTE Phase) (N=42) | Placebo-Riociguat (LTE Phase) (N=45) | Riociguat (Main Treatment Phase) (N=60) | Placebo (Main Treatment Phase) (N=61)
Palpitations (Cardiac disorders) | 3 (3) | 1 (1) | 8 (8) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 4 (6) | 4 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (3) | 2 (2) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (2) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (11) | 8 (23) | 10 (15) | 8 (11)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (3) | 7 (7) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (7) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 8 (8) | 15 (16) | 7 (7)
Nausea (Gastrointestinal disorders) | 2 (5) | 6 (7) | 7 (9) | 6 (6)
Vomiting (Gastrointestinal disorders) | 7 (11) | 4 (14) | 8 (14) | 6 (8)
Asthenia (General disorders) | 2 (2) | 1 (1) | 3 (6) | 3 (4)
Fatigue (General disorders) | 0 (0) | 4 (4) | 7 (7) | 6 (7)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 6 (7) | 2 (2)
Pain (General disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 5 (6) | 5 (5)
Bronchitis (Infections and infestations) | 5 (6) | 0 (0) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (13) | 10 (10) | 5 (7) | 5 (8)
Upper respiratory tract infection (Infections and infestations) | 7 (10) | 6 (7) | 4 (5) | 8 (10)
Urinary tract infection (Infections and infestations) | 2 (7) | 3 (4) | 4 (5) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (6) | 12 (14) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 4 (6) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3) | 4 (6) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 6 (7) | 13 (21) | 7 (7)
Headache (Nervous system disorders) | 3 (4) | 4 (4) | 11 (12) | 12 (16)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (5)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (4) | 9 (9) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4) | 8 (9) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (5) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (5) | 4 (4) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 5 (6) | 5 (9)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (4) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (4) | 4 (4) | 7 (9)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hypotension (Vascular disorders) | 5 (6) | 7 (9) | 7 (7) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 2 (2) | 3 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 5 (6) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 4 (5) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 1 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 1 (1) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any proposed publications should be sent to Bayer for review at least 40 days before forwarding to any person that is not bound by the confidentially obligations. Bayer may request delay of publication for no more than 120 days to allow for filing Patent Applications (if applicable). No publication of single center data should be done prior to publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT02283762/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT02283762/SAP_002.pdf